CLINICAL TRIAL: NCT04867382
Title: Reducing Stigma Toward People With Opioid Use Disorder Among Primary Care Clinicians
Brief Title: Comparing Two Training Methods for Opioid Wizard
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HealthPartners Institute (Other)
Collaborators: Hennepin Healthcare Research Institute (Other); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: A20-156; 3UG1DA040316-06S4 (NIH)
Record Dates: First submitted 2021-04-27; First posted 2021-04-30 (Actual); Results first posted 2022-12-15 (Actual); Last update posted 2022-12-15 (Actual); Status verified 2021-08

CONDITIONS: Opioid-use Disorder; Opioid Dependence; Attitude of Health Personnel
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Intervention Model Description: This study used a randomized controlled trial (RCT) design embedded in a larger, multisite trial of a clinical decision support (CDS) tool to help PCCs identify, diagnose, and treat patients with OUD. PCCs in clinics randomized to Opioid Wizard were randomized 1:1 to the intervention or comparison training and stratified by clinic.
Who Masked: Participant
Masking Description: Methods for concealment of allocation. PCCs were blind to their randomized MyLearning training assignment. The study statistician generated the randomization assignment, and a study team member submitted that list to HealthPartners (HP) MyLearning staff. Study team members collecting outcome data from surveys, Opioid Wizard, and Epic (including use rates, buprenorphine prescriptions) also were blinded to treatment assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): This arm received a case-based training on how to use the Opioid Wizard tool, including patient narratives and videos and person-first language.
  Interventions: Behavioral: Online training
- Comparison training (Placebo Comparator): This arm received a case-based training on how to use the Opioid Wizard tool.
  Interventions: Behavioral: Online training

INTERVENTIONS:
Behavioral: Online training — This intervention consisted of two different interactive online trainings delivered through an online learning platform at HealthPartners.

SUMMARY:
The prevalence of opioid use disorder (OUD) and opioid-related deaths has risen dramatically in recent years. Effective treatments, including medications for opioid use disorder (MOUDs; e.g., buprenorphine-naloxone and methadone) are under-utilized. There are few evidence-based interventions for changing attitudes toward Opioid Use Disorder (OUD) in the general public and especially among healthcare clinicians. This study proposed an innovative intervention to change attitudes of Primary Care Clinicians (PCCs) toward persons with OUD. Study participants were stratified into one of two online learning courses: the intervention training was compared with an attention-control training.

DETAILED DESCRIPTION:
Primary care offers an ideal setting in which to treat OUD; however, few clinicians are waivered to prescribe buprenorphine and of those who are waivered, less than one-third do prescribe. One potential barrier to increasing access to MOUDs are primary care clinician (PCC) attitudes towards people with OUD.

This study used a randomized controlled trial design to examine a novel intervention to change attitudes towards people with OUD among PCCs. PCCs in clinics randomized to the intervention in COMPUTE 2.0 (PCCs in 15 of the 30 clinics randomized in the parent study) were randomized 1:1 to the intervention or comparison training, stratified by clinic and waiver status. Training was conducted via MyLearning, an online learning software. All PCCs were asked to complete a brief training (25-35 minutes for both trainings) on the shared decision-making tool (SDM) called the Opioid Wizard, which alerts PCCs to screen, diagnose, and treat people with OUD. PCCs in the intervention arm heard patient narratives designed to shift attitudes about patients with OUD. PCCs in the comparison training had training on using the SDM tool. The PCCs were asked to complete a survey of attitudes and intentions to get waivered to prescribe buprenorphine immediately following the online training. Use of the CDS was monitored in both groups for 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Primary Care Clinician: Had to be a family physician, general internist, adult-care non-obstetric nurse practitioner, or a physician assistant
* Had to practice at a study-eligible primary care clinic already involved in the main study intervention arm

Exclusion Criteria:

PCCs were ineligible to participate if they had fewer than 5 eligible patient encounters between Sep 2020 and Feb 2021.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2021-04-09 (Actual); Primary Completion 2021-09-10 (Actual); Study Completion 2021-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Hooker, PhD, MPH, MS, Principal Investigator — HealthPartners Institute
Locations (1):
- HealthPartners, Bloomington, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Yes
As part of the HEAL initiative, the main study results, as described in the initial publication, will be shared on the HEAL Data Platform.
Time Frame: Pending
Access Criteria: You will not need to log in in order to: browse the study metadata on the Discovery Page or read the pre-made tutorial notebooks in the "Example Analysis" tab.
  You will need to log in and obtain authorization (access) in order to: register your own study; access studies with controlled data perform analyses in workspaces; and download data files and file manifests. run interactive tutorial notebooks in workspaces
URL: https://healdata.org/portal/discovery/3UG1DA040316-06S4/

REFERENCES:
- [Derived] Hooker SA, Crain AL, LaFrance AB, Kane S, Fokuo JK, Bart G, Rossom RC. A randomized controlled trial of an intervention to reduce stigma toward people with opioid use disorder among primary care clinicians. Addict Sci Clin Pract. 2023 Feb 11;18(1):10. doi: 10.1186/s13722-023-00366-1. PMID 36774521

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligible participants for this study were primary care providers (PCCs) who practice at HealthPartners Clinics that were previously randomized into the intervention arm of the parent study (NCT04198428). Family physician, general internist or adult-care non-obstetric nurse practitioner or physician assistant were the titles included. PCCs were eligible to participate regardless of whether they were waivered to prescribe buprenorphine. 162 PCCs were invited by email to participate in this study.
Pre-assignment Details: A total of 411 Primary Care Clinicians (PCCs) actively practicing at clinics within the parent study were screened for eligibility. They were ineligible to participate if:
  * They had fewer than 5 eligible patient encounters between Sep 2020 and Feb 2021 (N=50);
  * They practiced in a non-intervention clinic (n=199)
Groups:
- Intervention: The intervention arm received an online training in the use of the SDM tool that includes patient narratives and videos and person-first language.
- Comparison Training: The comparison training arm received an online training in the use of the SDM tool.
Period: Overall Study
Arm/Group | Intervention | Comparison Training
Started | 48 | 40
Completed Stigma Reduction (Intervention) or Attention-control (Comparison) Training | 48 | 40
Completed (Primary analysis conducted with data from those who completed survey immediately following the online training.) | 46 | 39
Not Completed | 2 | 1
Not completed — Did not complete the survey | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Intervention: The intervention arm received an online training in the use of the SDM tool that included patient narratives and videos and person-first language.
- Total: Total of all reporting groups
Arm/Group | Intervention | Comparison Training | Total
Number analyzed (Participants) | 48 | 40 | 88
Age, Categorical [Count of Participants; unit: Participants] — Population: Three participants completed the training but not the survey and we lack any demographic data on them.
  Participants
    number analyzed (Participants) | 46 | 39 | 85
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 40 | 34 | 74
    >=65 years | 6 | 5 | 11
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Three participants completed the training but not the survey and we lack any demographic data on them.
  years
    number analyzed (Participants) | 46 | 39 | 85
    (all) | 47.76 (11.85) | 47.00 (11.31) | 47.4 (11.6)
Sex/Gender, Customized [Count of Participants; unit: Participants] — Population: Three participants completed the training but not the survey and we lack any demographic data on them.
  Participants
    Male: number analyzed (Participants) | 46 | 39 | 85
    Male | 17 | 14 | 31
    Female: number analyzed (Participants) | 46 | 39 | 85
    Female | 27 | 22 | 49
    Not Listed: number analyzed (Participants) | 46 | 39 | 85
    Not Listed | 1 | 0 | 1
    Prefer not to answer: number analyzed (Participants) | 46 | 39 | 85
    Prefer not to answer | 1 | 3 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Three participants completed the training but not the survey and we lack any demographic data on them.
  Participants
    number analyzed (Participants) | 46 | 39 | 85
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 6 | 2 | 8
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 3 | 3 | 6
    White | 29 | 28 | 57
    More than one race | 1 | 1 | 2
    Unknown or Not Reported | 7 | 5 | 12
Region of Enrollment [Number; unit: participants]
  United States | 48 | 40 | 88
Waivered to prescribe buprenorphine [Count of Participants; unit: Participants] | 3 | 5 | 8
Type of provider degree [Count of Participants; unit: Participants] — Population: Three participants completed the training but not the survey and we lack any demographic data on them.
  Participants
    number analyzed (Participants) | 46 | 39 | 85
    Doctor of Medicine/Doctor of Osteopathic Medicine MD/DO | 30 | 25 | 55
    Physician Assistant/Nurse Practitioner PA/NP | 16 | 14 | 30

OUTCOME MEASURES:

1. Primary Outcome: Difference, Disdain, and Blame Scales
Description: Attitudes toward people with OUD were measured using the Difference, Disdain, and Blame scales, which measure attitudes toward people with mental illness and substance use disorders (SUDs). Difference, Disdain, and Blame scales measured stigma toward people with OUD, with three questions in each domain. Items are scored on a 9-point agreement scale. The range is 1-9; some items are reverse-scored. Items are averaged to obtain a score, with higher scores reflecting more stigma (range = 1-9). Evidence suggests that the scales demonstrate good internal consistency and are positively associated.
Time Frame: Immediately after completing online training.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Comparison Training
Number analyzed (Participants) | 46 | 39
score on a scale | 4.1 (1.3) | 4.3 (1.2)
Statistical Analysis 1: Comparison: Intervention vs Comparison Training; Test type: Superiority; p = .63, t-test, 2 sided; Mean Difference (Final Values) = -0.13, Standard Error of Mean 0.27

2. Secondary Outcome: Intentions to Get Waivered to Prescribe Buprenorphine.
Description: Non-waivered PCCs rated one question on their intention to get waivered to prescribe buprenorphine ("How likely are you to get waivered to prescribe buprenorphine in the next year?") on a five-point Likert-type scale ranging from 1 (I definitely will not) to 5 (I definitely will). Higher scores correspond to greater intention to get waivered.
Time Frame: Immediately after completing online training
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Comparison Training
Number analyzed (Participants) | 43 | 34
score on a scale | 2.3 (0.7) | 2.1 (0.8)
Statistical Analysis 1: Comparison: Intervention vs Comparison Training; Test type: Superiority; p = 0.27, t-test, 2 sided; Mean Difference (Final Values) = 0.19, Standard Error of Mean 0.17

3. Secondary Outcome: Intentions to Prescribe Buprenorphine Should a Waiver no Longer be Required.
Description: Non-waivered PCCs rated one question on their intentions to prescribe buprenorphine if a waiver were no longer required ("If your patient with OUD requested buprenorphine in the next year and a waiver were no longer required, would you prescribe buprenorphine?") on a five-point Likert-type scale ranging from 1 (I definitely would not) to 5 (I definitely would). Higher numbers indicate greater likelihood to prescribe buprenorphine.
Time Frame: Immediately after completing online training
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Comparison Training
Number analyzed (Participants) | 43 | 34
score on a scale | 3.2 (1.0) | 3.0 (0.9)
Statistical Analysis 1: Comparison: Intervention vs Comparison Training; Test type: Superiority; p = .37, t-test, 2 sided; Mean Difference (Final Values) = 0.20, Standard Error of Mean 0.22

4. Secondary Outcome: Opioid Wizard Use
Description: PCC Opioid Wizard use was defined as clicking within the tool, such as screening for OUD, making a diagnosis, providing a referral, prescribing a medication, printing patient education materials, or prescribing naloxone. This variable was dichotomized as whether the PCC ever clicked in the tool (1=yes; 0=no) in the 6 months following the training.
Time Frame: Six months following online training.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Comparison Training
Number analyzed (Participants) | 48 | 40
Participants | 3 | 4
Statistical Analysis 1: Comparison: Intervention vs Comparison Training; Test type: Superiority; p = .12, Regression, Logistic; Odds Ratio (OR) = 1.75, 95% CI 2-sided [0.86 to 3.57]

ADVERSE EVENTS:
Time Frame: Not collected.
Description: Adverse events were not monitored because this was a minimal-risk study.
Arm/Group | Intervention | Comparison Training
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
The online training meant there was no way for the research team to control for PCC engagement with content. The training, at 25-35 minutes, may not have been intensive enough to have substantial impact. The comparison training, which lasted the same amount of time and covered some of the same topics, may have had an effect on PCCs. The study did not include a baseline training to avoid signaling the primary outcome was stigma, so there is no way to measure pre-training attitudes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2021-11-23): https://cdn.clinicaltrials.gov/large-docs/82/NCT04867382/Prot_SAP_ICF_001.pdf